CLINICAL TRIAL: NCT05288361
Title: Determining the Cause of Coronary Vasomotor Disorders in Patients With Ischemia and No Obstructive Coronary Artery Disease
Brief Title: The DISCOVER INOCA Prospective Multi-center Registry
Acronym: DISCOVER INOCA
Status: Active, not recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: YSI-001
Record Dates: First submitted 2022-03-09; First posted 2022-03-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Ischemia and No Obstructive Coronary Artery Disease; Coronary Microvascular Dysfunction; Coronary Vasospasm; Endothelial Dysfunction; Microvascular Angina; Chest Pain With Normal Coronary Angiography
MeSH Terms: conditions — Ischemia; Coronary Vasospasm; Microvascular Angina

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Coroventis Coroflow Cardiovascular System and PressureWire™ X Guidewire — Patients presenting with symptomatic ischemic heart disease (including chronic stable angina or unstable angina) without evidence of myocardial infarction who require elective or urgent cardiac catheterization, and who meet all eligibility criteria will be enrolled.
  Participants will undergo routine coronary angiography as well as comprehensive physiologic assessment with intracoronary acetylcholine provocation for diagnosis of vasospastic angina (VSA), coronary thermodilution to evaluate for coronary microvascular dysfunction (CMD), and intracoronary imaging with optical coherence tomography (OCT) or intravascular ultrasound (IVUS) to evaluate for the presence of atheroma, plaque burden, and myocardial bridging.
  Other Names: Acetylcholine Provocation

SUMMARY:
The overall objective of this multi-center registry is to identify specific phenotypes of INOCA with both an anatomic evaluation (coronary angiography and intravascular imaging) and physiologic assessment with the Abbott Coroventis Coroflow Cardiovascular System, and to determine long-term outcomes.

DETAILED DESCRIPTION:
This is a prospective, multicenter, registry of stable patients with ischemia and no obstructive coronary artery disease (INOCA) evaluated by coronary angiography, intravascular imaging, and physiologic measurements obtained on the Coroventis Coroflow Cardiovascular System.

The Coroventis Coroflow Cardiovascular System and PressureWire™ X Guidewire (Abbott, Abbott Park, IL) are a device combination consisting of a physiology wire with wireless transmitter (Wi-Box), CoroHub Receiver, and CoroFlow Software. The PressureWire™ X guidewire is a hydrophilic-coated wire with pressure and temperature sensors that is capable of measuring physiologic indices including fractional flow reserve (FFR), resting full cycle ratio (RFR), coronary flow reserve (CFR), and the index of microcirculatory resistance (IMR). The guidewire wirelessly transmits pressure and temperature data via the Wi-Box to the CoroHub Receiver and CoroFlow Software, which is a software interface designed to display pressure measurements, thermodilution curves, and physiologic indices. This registry will enroll 500 subjects at up to 10 sites in the United States that use the Abbott Coroventis Coroflow Cardiovascular System.

The overall objective of this multi-center registry is to identify specific phenotypes of INOCA with both an anatomic evaluation (coronary angiography and intravascular imaging) and physiologic assessment with the Abbott Coroventis Coroflow Cardiovascular System, and to determine long-term outcomes. Specific goals include:

* Describe the prevalence of the following INOCA phenotypes: coronary microvascular dysfunction (CMD), vasospastic angina, mixed CMD/vasospastic angina, other disorders of coronary physiology, and non-cardiac chest pain;
* Characterize the burden of epicardial coronary artery atherosclerosis and myocardial bridging (MB) by angiography and intracoronary imaging (intravascular ultrasound or optical coherence tomography) in patients with INOCA;
* Characterize the natural history and outcomes of patients with INOCA and determine variables associated with major adverse cardiovascular events

ELIGIBILITY:
Inclusion Criteria:

* Suspected ischemic heart disease and is referred to undergo clinically indicated invasive coronary angiography
* No obstructive coronary artery disease (CAD) as defined by operator visual assessment with (1) angiographically normal coronary arteries OR (2) non-obstructive CAD with angiographic stenosis < 50%, or greater than or equal to 50 but < 70% with FFR greater than or equal to 0.81 or RFR greater than or equal to 0.90
* Willing to comply with specified follow-up evaluations. The participant or legally authorized representative has been informed of the nature of the study, agrees to its provisions, and has been provided written informed consent approved by the appropriate Institutional Review Board (IRB) or Ethics Committee (EC)

Exclusion Criteria:

* Pregnant or nursing
* Any myocardial infarction at index presentation or within 90 days prior to enrollment, defined as any electrocardiogram diagnostic for myocardial infarction OR elevation in serum troponin greater than the upper limit of the site-defined reference range
* Known left ventricular ejection fraction < 50% or cardiogenic shock requiring pressors or mechanical circulatory assistance (e.g., intra-aortic balloon pump, left ventricular assist device, other temporary cardiac support blood pump)
* Renal insufficiency, defined as estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2 (by the Modification of Diet in Renal Disease equation) or dialysis at the time of screening
* Prior percutaneous coronary intervention
* Planned percutaneous coronary intervention (PCI)
* Prior coronary artery bypass graft surgery
* Prior ST-elevation myocardial infarction
* History of hypertrophic cardiomyopathy
* History of infiltrative heart disease (e.g., cardiac amyloidosis)
* New York Heart Association Class IV congestive heart failure
* Severe mitral regurgitation
* Severe aortic stenosis
* Severe pulmonary hypertension (Mean pulmonary artery pressure greater than or equal to 35mmHg or echocardiographic right ventricular systolic pressure greater than or equal to 60mmHg)
* Known history of unrepaired or repaired congenital heart disease
* Past or pending heart transplant, or on the waiting list for organ transplant
* Known other medical illness or known history of substance abuse that may cause non-compliance with the protocol, or is associated with a life expectancy of less than 1 year
* Current or planned participation in a study of an investigational therapy
* Angiographic stenosis in any major epicardial vessel ≥ 70% by visual estimate
* Angiographic stenosis in any major epicardial vessel greater than or equal to 50% and < 70% by visual estimate with FFR less than or equal to 0.80 or RFR less than or equal to 0.89

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults referred to the catheterization laboratory for evaluation of suspected ischemic heart disease, and who are deemed to have non-obstructive coronary artery disease based on coronary angiography or non-ischemic fractional flow reserve (FFR) or resting free cycle ratio (RFR).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with each physiologic phenotypes diagnosed with the Coroflow Cardiovascular System will be reported within 24-48 hours of the procedure. | up to 48 hours after the procedure
  The following phenotypes will be captured: Coronary microvascular dysfunction (CMD)- Criteria for a diagnosis of CMD include an abnormal Index of Microcirculatory Resistance (IMR) ≥ 25 and/or impaired Coronary Flow Reserve (CFR) ≤ 2.0; Vasospastic angina (VSA): Includes coronary vasospasm, microvascular spasm, and endothelial dysfunction. Criteria for coronary vasospasm include ≥ 90% narrowing of the epicardial vessel during acetylcholine testing and either or both angina and transient ischemic EKG changes. Microvascular spasm includes angina and/or ischemic EKG changes in the absence of spasm of the epicardial vessel during acetycholine infusion; Endothelial dysfunction as defined as angiographic diameter change less than or equal to 0% and but not greater than -89% in response to acetylcholine infusion; Mixed CMD/VSA; Any other disorders of coronary physiology.
The proportion of subjects that experience Major Adverse Cardiovascular Events (MACE) | Up to 5 years
  The proportion of subjects that experience Major Adverse Cardiovascular Events (MACE) as reported by the clinical study sites and adjudicated by the Clinical Events Committee (CEC). Reports may come from the clinical site or self report. MACE defined as a composite of cardiovascular death, myocardial infarction, hospitalization for cardiovascular causes or coronary revascularization.
The proportion of subjects that exhibit mild, moderate or severe coronary artery stenosis | At the time of the procedure
  The proportion of subjects that exhibit mild, moderate or severe coronary artery stenosis as measured by Optical Coherence Tomography (OCT), Intravascular Ultrasound (IVUS) or Quantitative Coronary Angiography (QCA). Mild stenosis is defined as less than or equal to 30%, Moderate stenosis is defined as 31%-69%, and severe stenosis is greater than or equal to 70%. The measurements will take place during the procedure and the analysis will be completed by a central core lab.
Lesion length during the procedure | At the time of the procedure
  Lesion length during the procedure will be determined for each subject by the use of OCT, IVUS or QCA and the analysis will be completed by a central core lab. Lesion length will be defined by either less than 15mm or equal to or greater than 15mm.

SECONDARY OUTCOMES:
The proportion of subjects that experience Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) at any time during the study. | Up to 5 Years
  The proportion of subjects that experience Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) at any time during the study as reported by the clinical site or self report. MACCE is defined as MACE and/or any stroke (NeuroARC definition) and adjudicated by the CEC.
The proportion of subjects that die at any time in the study | Up to 5 years
  The proportion of subjects that die at any time in the study as reported by the clinical site or the subject's family. The cause of death will be further defined as cardiovascular, and non-cardiovascular mortality as adjudicated by the CEC.
The proportion of subjects that experience a Myocardial Infarction (MI) at any time during the study. | Up to 5 Years
  The proportion of subjects that experience a Myocardial Infarction (MI) at any time during the study as reported by the clinical site or self report. Fourth Universal Definition will be used to determine MI type and will be adjudicated by the CEC.
The proportion of subjects that experience a stroke at any time during the study. | Up to 5 years
  The proportion of subjects that experience a stroke at any time during the study as reported by the clinical site or self report. NeuroARC definition will be used to classify the type of stroke and will be adjudicated by the CEC.
The proportion of subjects that require revascularization of their coronary arteries at any time during the study. | Up to 5 years
  Reports may come from the clinical site or self report. Revascularization will further be defined as Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Graft (CABG) and will be adjudicated by the CEC.
The proportion of subjects that experience a hospitalization at any time during the study. | Up to 5 years
  The proportion of subjects that experience a hospitalization at any time during the study as reported by the clinical site or self report. The reason for hospitalization will be further classified as Cardiovascular related or Heart Failure and adjudicated by the CEC
The proportion of subjects that require repeat coronary angiography at any time during the study. | Up to 5 years
  The proportion of subjects that require repeat coronary angiography at any time during the study as reported by the clinical site or self report. Reported events will be adjudicated by the CEC.
The proportion of subjects with coronary lesions that experience progression to obstructive Coronary Artery Disease (CAD) at any time during the study. | Up to 5 years
  The proportion of subjects with coronary lesions that experience progression to obstructive Coronary Artery Disease (CAD) at any time during the study as reported by the clinical site or self report, and will be adjudicated by the CEC.
Proportion of subjects that experience major bleeding at any time during the study using the Bleeding Academic Research Consortium (BARC) bleeding type | Up to 5 years
  Proportion of subjects that experience major bleeding at any time during the study using the BARC bleeding type. Reports may come from the clinical site or self report. Bleeding types on a scale from 0 (no bleeding) to 5 (fatal bleeding). Major bleeding is defined as categories BARC 3-5 and will be adjudicated by the CEC.
Proportion of subjects that experience Major Vascular Complications at any time during the study. | Up to five 5 years
  Proportion of subjects that experience Major Vascular Complications at any time during the study as reports by the clinical site or self report, and will be adjudicated by the CEC.
Proportion of subjects that experience a composite of death, stroke, and MI at any time during the study. | Up to 5 years
  Proportion of subjects that experience a composite of death, stroke, and MI at any time during the study as reported by the clinical site or self report, and will be adjudicated by the CEC.
Change from baseline in proportion of subjects that experience each classification of angina status during the study. | At baseline, 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  The angina status will be assessed using the Canadian Cardiovascular Society (CCS) class or Braunwald Unstable Angina classification. The angina type will be classified at the time of the procedure, at 30 days, 6 months, 1 year, and then annually up to 5 years.
The change in baseline of angina symptoms for each subject. The angina status will be classified at the time of the procedure, at 30 days, 6 months, 12months and then annually up to 5 years. | At baseline, 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  The change in baseline of angina symptoms for each subject as assessed by the Seattle Angina Questionaire. The Seattle Angina Questionnaire (SAQ) contains 19 questions used to measure health status in patients with coronary artery disease (CAD). The SAQ directly measure patients' current health status: Physical Limitation, Angina Frequency, and Quality of Life. The SAQ results in 3 domain scores as well as an overall summary score.
The change in the quality of life (QOL) from baseline for each subject will be assessed using the QOL EQ-5D-5L questionnaire. | At baseline, 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  QOL will be assessed by EQ-5D-5L. The EQ-5D-5L consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).QOL will be determined at the time of the procedure, at 30 days, 6 months, 12months and then annually up to 5 years.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
The change in depression status from baseline for each subject assessed by the Patient Health Questionnaire (PHQ)-8 questionnaire. | At baseline, 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  Depression status will be assessed by the PHQ-8 questionnaire. The PHQ-8 is a series of 8 questions will four possible answers each. The questions focus on over-all well-being as well as daily habits. The higher the score the more the patient is likely to be depressed. Depression status will be determined at the time of the procedure, at 30 days, 6 months, 12months and then annually up to 5 years.
The change in anxiety status from baseline for each subject. will be assessed by the Generalized Anxiety Disorder (GAD)-7 questionnaire. | At baseline, 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years
  Anxiety status will be assessed by the GAD-7 questionnaire. The GAD-7 is a series of 7 questions will four possible answers each. The questions focus on over-all well-being as well as daily habits. The higher the score the more the patient is likely to be anxious. Anxiety status will be determined at the time of the procedure, at 30 days, 6 months, 12months and then annually up to 5 years.
The proportion of subjects that experience a series of procedural outcomes as assessed by the site and adjudicated by the CEC. | Up to 48 hours after the procedure
  Procedural outcomes will be categorized into the following: Reclassification from pre-procedure diagnosis (including non-cardiac chest pain); Completion of the interventional diagnostic procedure without device-related serious adverse events or major angiographic complications; Frequency of major angiographic complications (device-related coronary artery dissection [greater than type C], slow or no flow, or perforation)

CONTACTS AND LOCATIONS:
Overall Officials: Samit Shah, MD, PhD, Principal Investigator — Yale University Medical School; Alexandra Lansky, MD, Principal Investigator — Yale University Medical School
Locations (9):
- United States (9):
  - UCLA Health, Los Angeles, California
  - Stanford Hospital, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - New York Presbyterian-Brooklyn Methodist Hospital, Brooklyn, New York
  - NYU Langone Health, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No